CLINICAL TRIAL: NCT06809803
Title: Safety, Convenience, and Tolerability of a Nightly Single Oral Dose of Extended-release Sodium Oxybate in Children
Brief Title: Extended-release Sodium Oxybate in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Avadel (Industry)
Responsible Party: Principal Investigator, Oliver Sum-Ping, Clinical Associate Professor in Psych/Sleep Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 75896
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Narcolepsy Type 1 (NT 1)
Keywords: Narcolepsy; Children; Sodium oxybate; treatment
MeSH Terms: conditions — Narcolepsy | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Extended-release sodium oxybate (Experimental): Participants in this arm will take extended-release sodium oxybate
  Interventions: Drug: Extended-release sodium oxybate; Drug: Non-extended-release oxybates
- Non-extended-release oxybates (Active Comparator): Participants in this arm will take non-extended-release sodium oxybate
  Interventions: Drug: Extended-release sodium oxybate; Drug: Non-extended-release oxybates

INTERVENTIONS:
Drug: Extended-release sodium oxybate — Participants will take Extended-release sodium Oxybate (Lumryz) 4.5-9 g oral suspension in approximately ⅓ cup of water orally once a day before bedtime. Dosage of Lumryz will be the same as the equivalent total dose of the Non-Extended-release Oxybate (Xywav or Xyrem) that participants use before starting the study
  Other Names: Lumryz
Drug: Non-extended-release oxybates — Participants will take Non-Extended-release Oxybates (Xyrem oral solution or Xywav oral solution) 4.5-9 g orally per night (divided into two doses, once before bedtime and another dose 2-4 hours later) at the same dose of Xyrem or Xywav that participants use before starting the study will be continued to compare with Extended-release sodium Oxybate (Lumryz)
  Other Names: Xywav; Xyrem

SUMMARY:
The main objectives of this study are to determine the treatment preferences of children with narcolepsy type 1 between Extended-release sodium oxybate and Non-extended-release oxybates (Sodium oxybate or a medication with the combination of Calcium, magnesium, potassium, and sodium oxybates). The study will also assess the safety, convenience, and tolerability of Extended-release sodium oxybate. Additionally, the researchers aim to assess how well Extended-release sodium oxybate works in treating narcolepsy type 1.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be under the care of a doctor at the Stanford Sleep Clinic.
2. Participants must have a documented diagnosis of narcolepsy type 1 shown by sleepiness and either: a spinal fluid marker for narcolepsy (hypocretin-1) at a specific level, or a history of sudden loss of muscle control (cataplexy), or a particular genetic marker for narcolepsy, or a sleep study showing a specific sleep pattern for narcolepsy.
3. Parent(s), or guardian(s) have signed a consent form and the child must agree to participate.
4. Participants are on a stable dose of medications

Exclusion Criteria:

Participants who have any of the following conditions will not be included in the study

1. Uncontrolled mental health problems
2. Uncontrolled sleep problems that lead to sleepiness.
3. Currently having thought about ending one's life or sadness or loss of interest
4. Currently having a problem with illegal drug use
5. Currently pregnant

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Participant preference for selecting the extended vs non-extended release oxybates | Baseline, up to 8-12 weeks through study completion
  Participants will be asked at the end of the study whether participants prefer extended-release sodium oxybate vs sodium oxybate vs calcium, magnesium, potassium and sodium oxybates

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scales for Children and Adolescents (ESS-CHAD) score | Baseline, up to 8-12 weeks through study completion
  ESS-CHAD is a multi-item questionnaire which asks the participants to rate their chances of falling asleep during various normal daily activities. 4-point Likert scale will be used. The score ranges from 0-24. A higher score means higher chance of falling asleep.
Number of cataplexy attacks | Baseline, up to 8-12 weeks through study completion
  The study team will ask the participants to report the number of cataplexy attacks as measured by Sleep and Symptoms diary when participants switch to the other intervention.
Change in Patient Global Impression of Change (PGIc) scale score | Baseline, up to 8-12 weeks through study completion
  The PGIc is a 7-point scale. Participants will be asked to rate their narcolepsy impression since the end of the Stable-Dose Period. The scale is Very much better, Much better, A little better, No change, A little worse, Much worse, and Very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Sum-Ping, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No